CLINICAL TRIAL: NCT03657004
Title: Impact of Switch of Immunosuppressive Regime on Changes in Renal Function and Transplant Rejection Rate in Patients With Lung Transplant
Brief Title: Immunosuppressive Regimen on Changes in Renal Function and Transplant Rejection Rate in Patients With Lung Transplant
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Faeq Husain, Senior physician, University of Giessen
Other Study IDs: Giessen
Record Dates: First submitted 2018-08-29; First posted 2018-09-04 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-08

CONDITIONS: Lung Transplant; Complications; Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective single-center analyzes the impact of switch of immunosuppressive regimen on renal function and transplant rejection rate in patients with lung transplant.

DETAILED DESCRIPTION:
Lung transplantation (LTx) is the preferred treatment modality for patients with end-stage lung disease. However, despite significant advances in treatment after LTx, comorbidities and medical complications contribute to a major extend to the high morbidity and mortality rate. Chronic kidney disease is common in patients after lung transplantation, and a large proportion of these patients ultimately progress to end-stage renal disease requiring dialysis. Chronic calcineurin inhibitor nephrotoxicity is one of the major risk factors for the development of chronic kidney disease. Mammalian target of rapamycin (mTOR) inhibitors such as everolimus have been increasingly used in combination with calcineurin inhibitors to reduce nephrotoxicity. However, whether a mTOR inhibitor based immunosuppressive regime leads to lower chronic nephrotoxicity remains unknown. The aim of this study is to evaluate whether the switch of the standard immunosuppressive regime after LTx with mycophenolate/tacrolimus/prednisolon to everolimus/tacrolimus/prednisolon is associated with an improved long-term preservation of renal function without increase in rejection rate.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent lung transplantation at the University Hospital Giessen and Marburg, Campus Giessen and Kerckhoff Clinic Bad Nauheim

Exclusion Criteria:

* Patients who died within 3 months after lung transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent lung transplantation at the University Hospital Giessen and Marburg, Campus Giessen and Kerckhoff Clinic Bad Nauheim
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Long-term loss of renal function in patients with standard immunosuppressive regimen after LTx (mycophenolate/tacrolimus/prednisolon) compared to those who switch to a mammalian target of rapamycin inhibitor based immunosuppressive regime | 2003-2018
  Renal function as measured by estimated glomerular filtration rate (Chronic Kidney Disease Epidemiology Collaboration formula)

SECONDARY OUTCOMES:
Rates of rejection (acute and chronic) in patients with standard immunosuppressive regimen after LTx (mycophenolate/tacrolimus/prednisolon) compared to those who switch to a mammalian target of rapamycin inhibitor based immunosuppressive regime | 2003-2018
  Rejection as measured by histological assessment

CONTACTS AND LOCATIONS:
Overall Officials: Werner Seeger, MD, Study Director — University Hospital Giessen and Marburg, Department of Internal Medicine II
Locations (1):
- University Hospital Giessen and Marburg, Giessen, Hesse, Germany

REFERENCES:
- [Result] Hellemons ME, Bakker SJ, Postmus D, Verschuuren EA, Erasmus ME, Navis G, van der Bij W. Incidence of impaired renal function after lung transplantation. J Heart Lung Transplant. 2012 Mar;31(3):238-43. doi: 10.1016/j.healun.2011.08.013. Epub 2011 Oct 5. PMID 21975352
- [Result] Guethoff S, Stroeh K, Grinninger C, Koenig MA, Kleinert EC, Rieger A, Mayr T, von Ziegler F, Reichart B, Hagl C, Schramm R, Kaczmarek I, Meiser BM. De novo sirolimus with low-dose tacrolimus versus full-dose tacrolimus with mycophenolate mofetil after heart transplantation--8-year results. J Heart Lung Transplant. 2015 May;34(5):634-42. doi: 10.1016/j.healun.2014.11.025. Epub 2014 Dec 9. PMID 25701373